CLINICAL TRIAL: NCT03850782
Title: A Phase 3b Study to Evaluate the Duration of Effect of Bimatoprost SR in Participants With Open-Angle Glaucoma or Ocular Hypertension
Brief Title: Evaluation of the Duration of Effect of Bimatoprost SR in Participants With Open-Angle Glaucoma or Ocular Hypertension
Acronym: TRITON
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1698-301-007; 2018-002574-52 (EudraCT Number); 2022-502380-37-00 (Other: EU CT)
Expanded Access: NCT05338606 (No longer available)
Record Dates: First submitted 2019-02-11; First posted 2019-02-22 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Open-Angle Glaucoma; Ocular Hypertension
Keywords: Open-Angle Glaucoma (OAG); Ocular Hypertension (OHT); Bimatoprost
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Bimatoprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bimatoprost SR - Dose A (Experimental): Study Eye: Participants will receive 1 - 2 Cycles of Bimatoprost SR administrations of Dose A
  Fellow Eye: The eye that does not receive Bimatoprost SR treatment will receive standard of care or up to one administration of Bimatoprost SR.
  Interventions: Drug: Bimatoprost (SR)
- Bimatoprost SR - Dose B (Experimental): Study Eye: Participants received 1 - 3 Cycles of Bimatoprost SR administrations of Dose B
  Fellow Eye: The eye that does not receive Bimatoprost SR treatment will receive standard of care or up to one administration of Bimatoprost SR.
  Interventions: Drug: Bimatoprost (SR)

INTERVENTIONS:
Drug: Bimatoprost (SR) — Study Eye: Cycles 1 - 3 administrations through the PRN treatment period.
  Fellow Eye: Standard of care or Bimatoprost SR.

SUMMARY:
This study evaluates the duration of intraocular pressure (IOP)-lowering effect and safety of as needed administrations of Bimatoprost sustained release (SR) in participants with open-angle glaucoma (OAG) or ocular hypertension (OHT) who are not adequately managed with topical IOP-lowering medication for reasons other than medication efficacy.

ELIGIBILITY:
Inclusion Criteria:

- Diagnosis of either open angle glaucoma (OAG) (i.e., primary OAG, pseudoexfoliation glaucoma, pigmentary glaucoma) or ocular hypertension requiring intraocular pressure-lowering treatment.

Exclusion Criteria:

* Concurrent or anticipated enrollment in another investigational drug or device study or participation in such a study within 2 months prior to enrolling in this study.
* Previous administration with Bimatoprost SR in the study eye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 515 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2025-08-08 (Actual); Study Completion 2025-08-08 (Actual)

PRIMARY OUTCOMES:
Retreatment or rescue administered for IOP | Up to 48 months
  Treatment modality determined by investigator.
Number of patients experiencing a treatment emergent adverse event | Baseline up to 48 months
  The number of patients who experienced one or more TEAE during the 48 month treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (108):
- United States (38):
  - Horizon Eye Specialists & Lasik Centers /ID# 235240, Sun City, Arizona
  - Atlantis Eye Care /ID# 235530, Huntington Beach, California
  - Lakeside Vision Center /ID# 234970, Irvine, California
  - Global Research Foundation /ID# 237350, Los Angeles, California
  - The Eye Research Foundation /ID# 234521, Newport Beach, California
  - Byers Eye Institute Stanford /ID# 235544, Palo Alto, California
  - Foothill Eye Institute /ID# 235640, Pasadena, California
  - Connecticut Eye Consultants P.C. /ID# 234981, Danbury, Connecticut
  - Advanced Research, LLC /ID# 236045, Deerfield Beach, Florida
  - Segal Drug Trials, Inc /ID# 235784, Delray Beach, Florida
  - International Research Center /ID# 238050, Tampa, Florida
  - Thomas Eye Group PC /ID# 235737, Sandy Springs, Georgia
  - Indiana University - Glick Eye Institute /ID# 235886, Indianapolis, Indiana
  - Retina Partners Midwest, PC /ID# 237876, Indianapolis, Indiana
  - Tulane University School of Medicine /ID# 237632, New Orleans, Louisiana
  - Ophthalmic Consultants of Boston /ID# 236534, Boston, Massachusetts
  - Clinical Eye Research of Boston LLC /ID# 234966, Winchester, Massachusetts
  - University of Michigan, Kellogg Eye Center /ID# 236496, Ann Arbor, Michigan
  - Fraser Eye Center /ID# 235790, Fraser, Michigan
  - Silverstein Eye Centers /ID# 237881, Kansas City, Missouri
  - Moyes Eye Centers /ID# 234989, Kansas City, Missouri
  - Alterman Modi & Wolter /ID# 235248, Poughkeepsie, New York
  - The Ohio State University /ID# 236790, Columbus, Ohio
  - AMA Eyes Research Institute /ID# 235542, Marysville, Ohio
  - Dean McGee Eye Institute /ID# 236823, Oklahoma City, Oklahoma
  - Oklahoma Eye Surgeons /ID# 235849, Oklahoma City, Oklahoma
  - Drs Fine Hoffman & Sims LLC /ID# 235918, Eugene, Oregon
  - Ophthalmic Partners, PC /ID# 235741, Bala-Cynwyd, Pennsylvania
  - Scott and Christie and Associates /ID# 234593, Cranberry Township, Pennsylvania
  - Black Hills Regional Eye Institute /ID# 235075, Rapid City, South Dakota
  - Vance Thompson Vision /ID# 235072, Sioux Falls, South Dakota
  - Eye Specialty Group /ID# 235721, Memphis, Tennessee
  - Vanderbilt University Medical Center /ID# 237177, Nashville, Tennessee
  - Advancing Vision Research /ID# 236681, Smyrna, Tennessee
  - ATX Clinical Trials Inc. dba Keystone Research /ID# 235868, Austin, Texas
  - Medical Center Ophthalmology Associates - Keystone Research /ID# 235787, San Antonio, Texas
  - Southern Utah Medical Research /ID# 235602, St. George, Utah
  - Piedmont Eye Center /ID# 234534, Lynchburg, Virginia
- Argentina (7):
  - Consultorio Oftalmologico Dr. Fabian Lerner /ID# 235855, CABA, Buenos Aires
  - Hospital Universitario Austral /ID# 237727, Pilar, Buenos Aires
  - Centro oftalmologico Dr Charles /ID# 235881, Ciudad de Buenos Aires, Buenos Aires F.D.
  - Oftalmología Global /ID# 239187, Rosario, Santa Fe Province
  - Hospital Italiano /ID# 235851, Buenos Aires
  - Centro Privado de Ojos /ID# 241283, Ciudad Autonoma Buenos Aires
  - Oftar Mendoza /ID# 240535, Mendoza
- Eye Surgery Associates /ID# 235873, East Melbourne, Victoria, Australia
- Bulgaria (14):
  - Multiprofile Hospital for Active Treatment "Lozenetz" /ID# 244053, Sofiya, Sofia
  - Diagnostic Consultative Center Aleksandrovska /ID# 238105, Sofiya, Sofia
  - Medical Center Oxycom Burgas /ID# 235580, Burgas
  - UMHAT Sveti Georgi /ID# 237027, Plovdiv
  - MHAT Hadzhi Dimitar /ID# 238248, Sliven
  - MHAT Dr. Bratan Shukerov /ID# 235498, Smolyan
  - Medical center for eye healt Focus Ltd /ID# 235575, Sofia
  - Pentagram Eye Hospital /ID# 235813, Sofia
  - Specialized Hospital for Active Treatment in Ocular Diseases "Zrenie" /ID# 235500, Sofia
  - St. Sofia Hospital /ID# 235525, Sofia
  - Medical Center -Verea /ID# 235494, Stara Zagora
  - Medical center Orfey /ID# 237344, Stara Zagora
  - MHAT Trakia /ID# 238137, Stara Zagora
  - Specialized Ophthalmological Hospital for Active Treatment - Varna /ID# 235962, Varna
- Czechia (3):
  - Všeobecná Fakultní Nemocnice v Praze /ID# 234422, Prague, Praha 17
  - Ocni klinika Pardubice /ID# 235944, Pardubice
  - Fakultni nemocnice Kralovske Vinohrady /ID# 234323, Prague
- Rigshospitalet Glostrup /ID# 235743, Glostrup Municipality, Capital Region, Denmark
- Germany (9):
  - Universitatsklinikum Freiburg /ID# 238048, Freiburg im Breisgau, Baden-Wurttemberg
  - Universitaetsmedizin Goettingen /ID# 237377, Göttingen, Lower Saxony
  - Universitaetsmedizin Rostock /ID# 237263, Rostock, Mecklenburg-Vorpommern
  - Universitaetsklinikum Schleswig-Holstein Campus Kiel /ID# 237069, Kiel, Schleswig-Holstein
  - Klinikum Dresden Friedrichstadt /ID# 235308, Dresden
  - Asklepios Kinik Nord - Heidberg Augenklinik /ID# 235955, Hamburg
  - St. Franziskus-Hospital /ID# 237714, Münster
  - Dietrich-Bonhoeffer-Klinikum /ID# 235262, Neubrandenburg
  - Augenzentrum Dr Hamacher /ID# 235537, Starnberg
- Hungary (4):
  - Gyongyosi Bugat Pal Korhaz /ID# 238144, Gyöngyös, Heves County
  - Vas Varmegyei Markusovszky Egyetemi Oktatokorhaz /ID# 237383, Szombathely, Vas County
  - Budapest Retina Intezet /ID# 235950, Budapest
  - Jahn Ferenc Del-pesti Korhaz es Rendelointezet /ID# 237111, Budapest
- Ireland (2):
  - Royal Victoria Eye and Ear Hospital /ID# 235546, Dublin
  - Institute of Eye Surgery /ID# 235547, Waterford
- Italy (7):
  - University of Catanzaro /ID# 238066, Catanzaro, Calabria
  - Sapienza University of Rome - Polo Pontino /ID# 237451, Terracina, Latina
  - Duplicate_Eye Clinic University of Catania /ID# 235573, Catania
  - Duplicate_Ospedale Ss. Annunziata /ID# 236587, Chieti
  - Fondazione IRCCS Policlinico San Matteo /ID# 236909, Pavia
  - University of Perugia /ID# 235811, Perugia
  - Fondazione Bietti - Ospedale Britannico /ID# 235495, Rome
- New Zealand (2):
  - Southern Eye Specialists /ID# 236080, Christchurch, Canterbury
  - Capital Eye Specialists /ID# 236112, Wellington
- Poland (5):
  - Wojskowy Instytut Medyczny /ID# 237031, Warsaw, Masovian Voivodeship
  - Optimum Profesorskie Centrum Okulistyki SP.z.o.o. /ID# 237076, Gdansk, Pomeranian Voivodeship
  - Centrum Diagnostyki i Mikrochirurgii Oka - LENS sp. z o.o /ID# 235928, Olsztyn, Warmian-Masurian Voivodeship
  - Gabinet Okulistyczny Edward Wylegala /ID# 235946, Katowice
  - Medical Center Julianow /ID# 235961, Lodz, Łódź Voivodeship
- S. Fyodorov Eye Microsurgery Federal State Institution /ID# 235984, Novosibirsk, Novosibirsk Oblast, Russia
- South Africa (2):
  - Pretoria Eye Institute - Private Practice /ID# 235658, Pretoria, Gauteng
  - Somerset Eye Specialist Medical & Surgical Centre /ID# 235540, Somerset West, Western Cape
- Norrlands University hospital /ID# 237553, Umeå, Västerbotten County, Sweden
- United Kingdom (11):
  - Addenbrookes Hospital /ID# 238255, Cambridge, Cambridgeshire
  - Mid Essex Hospitals NHS Trust /ID# 237776, Chelmsford, Essex
  - The Princess Alexandra NHS Trust /ID# 234433, Harlow, Essex
  - Kings College Hospital NHS Foundation Trust /ID# 237275, London, Greater London
  - York Hospital /ID# 237683, York, North Yorkshire
  - Oxford University Hospitals NHS Foundation Trust /ID# 237282, Oxford, Oxfordshire
  - East Suffolk and North Essex NHS Foundation Trust /ID# 234657, Colchester
  - Mid-Cheshire Hospitals NHS Trust /ID# 235418, Crewe
  - Liverpool University Hospitals NHS Foundation Trust /ID# 237095, Liverpool
  - Liverpool University Hospitals NHS Foundation Trust /ID# 237321, Liverpool
  - Central Middlesex Hospital /ID# 236216, London

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Silverstein SM, Oddone F, Kolko M, Brinkmann CK, Christie WC, Bicket AK, Gous PNJ, Luebke J, Maram J, Nguyen A, Craven ER, Pu Y, Jiao J, Bejanian M, Robinson MR; TRITON Study Group. Safety and Longevity of Intraocular Pressure Control After Bimatoprost Implant Administration: Interim Analysis of a Phase 3b Clinical Trial (TRITON). Drugs. 2025 Apr;85(4):557-570. doi: 10.1007/s40265-025-02154-4. Epub 2025 Feb 22. PMID 39985740
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=1698-301-007